CLINICAL TRIAL: NCT00501007
Title: Predictors of Treatment Outcome for Smokers With and Without Schizophrenia
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marc L. Steinberg, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: K23DA018203 (NIH); K23DA018203 (NIH)
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-psychiatric smokers: Smokers not meeting criteria for Schizophrenia or Schizoaffective Disorder
- Smokers with Schizophrenia: Smokers meeting criteria for schizophrenia or schizoaffective disorder

SUMMARY:
The primary purpose of this investigation is to determine the predictive value of task persistence as measured by a mirror tracing task. A secondary purpose is to evaluate differences in task persistence in smokers with or without schizophrenia. It is hypothesized that task persistence in smokers in both diagnostic categories (schizophrenia and no schizophrenia) will predict tobacco dependence treatment outcome at one and six months. It is also hypothesized that smokers with schizophrenia will show lower levels of task persistence after controlling for other motor skills than smokers without schizophrenia.

DETAILED DESCRIPTION:
Please see brief summary above.

ELIGIBILITY:
Inclusion Criteria:

* Current smokers must be over the age of 18,
* Must fit into the diagnostic groups schizophrenia / schizoaffective disorder; or the non-schizophrenia group.
* Must smoke at least 10 cigarettes per day
* Must be capable of giving informed consent as measured by Folstein Mini Mental Status Exam of at least 22.

Exclusion Criteria:

* Those unable to give informed consent.
* Psychotic disorders other than schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals from mental health centers in Central New Jersey or non-psychiatric controls from the community
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2005-02; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc L. Steinberg, PH.D, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ Tobacco Dependence Clinic, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 203 smokers were recruited from New Jersey state funded tobacco dependence treatment clinics, called QuitCenters, through clinician referrals or responses to recruitment flyers.
Pre-assignment Details: Reasons for exclusion included the following: Failed diagnostic screen, passed quit date/already using smoking cessation medications, changed mind about participating, smoked fewer than 10 cigarettes per day, did not have a goal to quit smoking, transportation issues, lost contact before baseline appointment, and low mini Mental Status Exam score.
Groups:
- Non-psychiatric Smokers: Smokers without a diagnosis of schizophrenia or schizoaffective disorder
- Smokers With Schizophrenia / Schizoaffective Disorder: Smokers meeting criteria for schizophrenia or schizoaffective disorder
Period: Overall Study
Arm/Group | Non-psychiatric Smokers | Smokers With Schizophrenia / Schizoaffective Disorder
Started | 100 | 103
Completed | 71 | 78
Not Completed | 29 | 25
Not completed — Inclusion criteria not met. | 29 | 25

BASELINE CHARACTERISTICS:
Groups:
- Diagnosis: Non-psychiatric group vs. Schizophrenia / Schizoaffective disorder
Arm/Group | Diagnosis
Number analyzed (Participants) | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 203
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.12 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 110
Region of Enrollment [Number; unit: participants]
  United States | 203

OUTCOME MEASURES:

1. Primary Outcome: Mirror-tracing Persistence (in Seconds)
Description: Number of seconds participants continued working on a mirror tracing task before giving up.
Time Frame: baseline
Population: All meeting inclusion criteria
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Schizophrenia or Schizoaffective Disorder: Smokers meeting Diagnostic and Statistical Manual criteria for Schizophrenia or Schizoaffective Disorder
- Non-psychiatric Group: Smokers NOT meeting criteria for schizophrenia, schizophrenia, bipolar disorder.
Arm/Group | Schizophrenia or Schizoaffective Disorder | Non-psychiatric Group
Number analyzed (Participants) | 78 | 71
seconds | 61.08 (57.38) | 100.34 (73.23)

2. Secondary Outcome: Persistence as a Prospective Predictor of Smoking Cessation
Description: Analysis of Generalized Estimating Equations (GEE) parameter estimates based on empirical standard error estimates, using an exchangeable working correlation structure, with smoking abstinence as outcome variable, and task persistence, time, diagnosis, ability, Fagerstrom Test for Nicotine Dependence (FTND) score, and the interaction between disorder and persistence as explanatory variables.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Odds ratio
Groups:
- Smoking Cessation: Participants received tobacco dependence treatment
Arm/Group | Smoking Cessation
Number analyzed (Participants) | 149
Odds ratio | 1.014 [1.014 to 1.017]

ADVERSE EVENTS:
Description: No adverse events were reported by participants to investigators during this study.
Arm/Group | Diagnosis
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes